CLINICAL TRIAL: NCT01691508
Title: MEA115575: A Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study of Mepolizumab Adjunctive Therapy to Reduce Steroid Use in Subjects With Severe Refractory Asthma
Brief Title: Mepolizumab Steroid-Sparing Study in Subjects With Severe Refractory Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115575
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Safety; Steroid Reduction; Efficacy; SB-240563; Eosinophils; Quality of Life; Mepolizumab; Severe Refractory Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mepolizumab (Experimental): Mepolizumab 100 mg subcutaneous once every 4 weeks upto Week 20
  Interventions: Drug: Mepolizumab; Drug: OCS (prednisone/prednisolone)
- Placebo (Experimental): Placebo subcutaneous once every 4 weeks upto Week 20
  Interventions: Drug: Placebo; Drug: OCS (prednisone/prednisolone)

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab is a fully humanised Immunoglobulin G antibody (IgG1, kappa) with human heavy and light chain frameworks.
  Arms: Mepolizumab
Drug: Placebo — Will be available as an equivalent volume of 0.9% sodium chloride.
  Arms: Placebo
Drug: OCS (prednisone/prednisolone) — Oral Corticosteroid (prednisone/prednisolone)

SUMMARY:
This is a randomised, double-blind, placebo-controlled, parallel-group, multicenter study of mepolizumab in comparison with placebo in reducing Oral Corticosteroid (OCS) use in subjects with severe refractory asthma. The study consists of four phases, OCS Optimisation Phase (Week -8 to Week 0), and the double-blind treatment period divided into an Induction Phase (Week 0 to Week 4), OCS Reduction Phase (Week 5 upto Week 20) followed by Maintenance Phase (Week 20 to Week 24). During the Optimisation Phase the investigator will adjust the OCS (prednisone/prednisolone) dose according to the Optimisation titration schedule based on a review of Asthma Control Questionnaire (ACQ)-5 score and exacerbation. In the Induction Phase subjects will be randomized 1:1 (approximately 60 per arm) to receive either mepolizumab (100 mg) administered subcutaneously (SC) or placebo every 4 weeks in addition to their existing maintenance asthma therapy with the lowest dose of OCS from Optimisation Phase. The Induction Phase will allow sufficient time for those subjects randomised to the mepolizumab arm to achieve a decrease in the eosinophilic inflammation prior to the reduction in OCS. During the Reduction Phase, subjects will continue receiving 100 mg mepolizumab/placebo every 4 weeks and the OCS dose reduction will be done every 4 weeks using the reduction titration schedule based on a review of eDiary parameters recorded by the subject, the subjects' exacerbation history, and a review of the signs and symptoms of adrenal insufficiency. In the Maintenance Phase subjects will be maintained without any further OCS dose adjustment. Subjects who complete the 24 week double-blind period and meet the eligibility criteria, will be offered the opportunity to participate in an open label extension (OLE) study otherwise they will return for a Follow-up Visit 12 weeks after their last dose of double blind study treatment. At each clinic visit, adverse events, safety labs, spirometery parameters and exacerbations will be assessed. The pharmacokinetic samples will be collected in the beginning of the treatment, prior to last dose, at the end of study (exit visit) and the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent and Study Compliance: Subjects must be able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form.
* Systemic Corticosteroids: Requirement for regular treatment with maintenance systemic corticosteroids in the 6 months prior to Visit 1 and using a stable oral corticosteroid dose for 4 weeks prior to Visit 1. Subjects must be taking 5.0 to 35 mg/day of prednisone or equivalent at Visit 1 and must agree to switch to study required prednisone/prednisolone as their oral corticosteroid and use it per protocol for the duration of the study.
* Inhaled Corticosteroids: Requirement for regular treatment with high dose inhaled corticosteroid in the 6 months prior to Visit 1. For 18 years of age and older: inhaled corticosteroid (ICS) dose must be >=880 microgram (µg)/day fluticasone propionate (FP) (ex-actuator) or equivalent daily. For ICS/ long acting beta2 agonist (LABA) combination preparations, the highest approved maintenance dose in the local country will meet this ICS criterion. For ages 12 to 17: ICS dose must be >=440 μg/day FP (ex-actuator) or equivalent daily.
* Controller Medication: Current treatment with an additional controller medication for at least 3 months OR documentation of having used and failed an additional controller medication for at least 3 successive months during the prior 12 months [e.g., LABA, leukotriene receptor antagonist (LTRA), or theophylline].
* Eosinophilic Asthma: Prior documentation of eosinophilic asthma or high likelihood of eosinophilic asthma.
* FEV1: Persistent airflow obstruction as indicated by a pre-bronchodilator FEV1 <80% predicted.
* Asthma: Evidence of asthma indicated by airway reversibility, hyperresponsiveness or airway variability.

Exclusion Criteria:

* Smoking history: Current smokers or former smokers with a smoking history of >=10 pack years.
* Concurrent Respiratory Disease: Presence of a clinically important lung condition other than asthma.
* Malignancy: A current malignancy or previous history of cancer in remission for less than 12 months prior screening
* Liver Disease: Unstable liver disease
* Cardiovascular: Subjects who have severe or clinically significant cardiovascular disease uncontrolled with standard treatment.
* Other Concurrent Medical Conditions: Subjects who have known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
* Eosinophilic Diseases: Subjects with other conditions that could lead to elevated eosinophils such as Hypereosiniophilic Syndromes, including Churg-Strauss Syndrome, or Eosinophilic Esophaghitis. Subjects with a known, pre-existing parasitic infestation within 6 months prior to Visit 1 are also to be excluded.
* ECG: ECG assessment QTcF >=450 milliseconds (msec) or QTcF >= 480 msec for subjects with Bundle Branch Block.
* Immunodeficiency: A known immunodeficiency (e.g. human immunodeficiency virus - HIV), other than that explained by the use of corticosteroids taken as therapy for asthma.
* Omalizumab Use: Subjects who have received omalizumab [Xolair] within 130 days of Visit 1.
* Other Monoclonal Antibodies: Subjects who have received any monoclonal antibody (other than Xolair) to treat inflammatory disease within 5 half-lives of Visit 1.
* Investigational Medications: Subjects who have received treatment with an investigational drug within the past 30 days or five terminal phase half-lives of the drug whichever is longer, prior to Visit 1 (this also includes investigational formulations of marketed products).
* Hypersensitivity: Subjects with a known allergy or intolerance to a monoclonal antibody or biologic.
* Pregnancy: Subjects who are pregnant or breastfeeding. Patients should not be enrolled if they plan to become pregnant during the time of study participation.
* Alcohol/Substance Abuse: A history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Visit 1.
* Adherence: Subjects who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations.
* Previous participation: Subjects who have previously any study of mepolizumab and received Investigational Product.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (44):
- United States (8):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Spartanburg, South Carolina
- Australia (4):
  - GSK Investigational Site, New Lambton, New South Wales
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (3):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- France (5):
  - GSK Investigational Site, Gières
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
- Germany (9):
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
- Mexico (2):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Rotterdam
- Poland (3):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
- United Kingdom (4):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Casale TB, Burnette A, Bourdin A, Howarth P, Hahn B, Stach-Klysh A, Khurana S. Oral corticosteroid-sparing effects of mepolizumab in severe eosinophilic asthma: evidence from randomized controlled trials and real-world studies. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107313. doi: 10.1177/17534666221107313. PMID 35972211
- [Derived] Khurana S, Brusselle GG, Bel EH, FitzGerald JM, Masoli M, Korn S, Kato M, Albers FC, Bradford ES, Gilson MJ, Price RG, Humbert M. Long-term Safety and Clinical Benefit of Mepolizumab in Patients With the Most Severe Eosinophilic Asthma: The COSMEX Study. Clin Ther. 2019 Oct;41(10):2041-2056.e5. doi: 10.1016/j.clinthera.2019.07.007. Epub 2019 Aug 22. PMID 31447130
- [Derived] Yancey SW, Bradford ES, Keene ON. Disease burden and efficacy of mepolizumab in patients with severe asthma and blood eosinophil counts of >/=150-300 cells/muL. Respir Med. 2019 May;151:139-141. doi: 10.1016/j.rmed.2019.04.008. Epub 2019 Apr 8. PMID 31047111
- [Derived] Ortega HG, Meyer E, Brusselle G, Asano K, Prazma CM, Albers FC, Mallett SA, Yancey SW, Gleich GJ. Update on immunogenicity in severe asthma: Experience with mepolizumab. J Allergy Clin Immunol Pract. 2019 Sep-Oct;7(7):2469-2475.e1. doi: 10.1016/j.jaip.2019.03.042. Epub 2019 Apr 5. No abstract available. PMID 30954640
- [Derived] Keene ON. Strategies for composite estimands in confirmatory clinical trials: Examples from trials in nasal polyps and steroid reduction. Pharm Stat. 2019 Jan;18(1):78-84. doi: 10.1002/pst.1909. Epub 2018 Oct 29. PMID 30370691
- [Derived] Magnan A, Bourdin A, Prazma CM, Albers FC, Price RG, Yancey SW, Ortega H. Treatment response with mepolizumab in severe eosinophilic asthma patients with previous omalizumab treatment. Allergy. 2016 Sep;71(9):1335-44. doi: 10.1111/all.12914. Epub 2016 May 24. PMID 27087007
- [Derived] Bel EH, Wenzel SE, Thompson PJ, Prazma CM, Keene ON, Yancey SW, Ortega HG, Pavord ID; SIRIUS Investigators. Oral glucocorticoid-sparing effect of mepolizumab in eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1189-97. doi: 10.1056/NEJMoa1403291. Epub 2014 Sep 8. PMID 25199060
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted 4 phases: oral corticosteroids (OCS) Optimization (Run-in); Induction; OCS Reduction and Maintenance. Participants (par.) who completed the 4 phases and met the eligibility criteria were offered the opportunity to participate in an open label extension (OLE) study. Par. not entering the OLE study completed the Follow-up Visit.
Pre-assignment Details: A total of 185 par. were screened; 3 par. were Screen failures; 47 par. were Run-in failures; 135 par. were randomized and received >=1 dose of study drug.
Groups:
- Placebo: Participants received placebo subcutaneously (SC) every 4 weeks (for a total of 6 doses),with the last dose at Week 20. A topical anaesthetic was permitted at the injection site to minimize discomfort, as needed. Rescue personnel and rescue medications (salbutamol/albuterol) /equipment were available throughout the study.
- Mepolizumab 100mg SC: Participants received mepolizumab 100 mg SC every 4 weeks (for a total of 6 doses), with the last dose at Week 20. A topical anaesthetic was permitted at the injection site to minimize discomfort, as needed. Rescue personnel and rescue medications (salbutamol/albuterol) /equipment were available throughout the study.
Period: Overall Study
Arm/Group | Placebo | Mepolizumab 100mg SC
Started | 66 | 69
Completed | 62 | 66
Not Completed | 4 | 3
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mepolizumab 100 mg SC: Participants received mepolizumab 100 mg SC every 4 weeks (for a total of 6 doses), with the last dose at Week 20. A topical anaesthetic was permitted at the injection site to minimize discomfort, as needed. Rescue personnel and rescue medications (salbutamol/albuterol) /equipment were available throughout the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Mepolizumab 100 mg SC | Total
Number analyzed (Participants) | 66 | 69 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (10.30) | 49.8 (14.10) | 49.9 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 44 | 74
  Male | 36 | 25 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian - Central/South Asian Heritage | 1 | 0 | 1
  Asian - East Asian Heritage | 0 | 1 | 1
  Asian - South East Asian Heritage | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White - Arabic/North African Heritage | 1 | 2 | 3
  White - White/Caucasian/European Heritage | 60 | 65 | 125
  Mixed Race | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Percent Reduction From Baseline in Oral Corticosteroid (OCS) Dose During Weeks 20 to 24 While Maintaining Asthma Control
Description: Baseline (BL) dose was the prescribed optimized prednisone/prednisolone dose following the OCS Optimization Phase. Maintenance (MN) dose was the mean of all daily prednisone/prednisolone doses during the MN Phase (weeks 20 to 24). The percent reduction of OCS dose during weeks 20 to 24 compared to BL dose was calculated as: 100 x (BL dose minus MN dose)/BL dose. Asthma control between weeks 20 and 24 was defined as no clinically significant exacerbation (worsening of asthma that required use of systemic corticosteroids or hospitalization and/or emergency department visits) during this period. The percent reduction of OCS was categorized as: 90 to 100%; 75 to <90%; 50 to <75%; >0 to <50%; no decrease in prednisone dose, or lack of asthma control, or withdrawal (WD) from treatment. Analysis was performed using a proportional odds model with terms for treatment group, region, duration of OCS use at BL (<5 years vs. >=5 years) and BL OCS dose.
Time Frame: Baseline; Weeks 20 to 24
Population: Intent-to-Treat (ITT) Population: all participants who were randomized and who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 66 | 69
Participants
  90 to 100% | 7 | 16
  75 to <90% | 5 | 12
  50 to <75% | 10 | 9
  >0 to <50% | 7 | 7
  No decrease /lack of asthma control/early WD | 37 | 25
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority or Other; p = 0.008, Proportional odds model; Odds Ratio (OR) = 2.39, 95% CI 2-sided [1.25 to 4.56]

2. Secondary Outcome: Number of Participants Who Achieved a Reduction of >=50% in Their Daily Oral Corticosteroid (OCS) Dose Compared With Baseline Dose, During Weeks 20 to 24 While Maintaining Asthma Control
Description: Baseline (BL) dose was the prescribed optimized prednisone/prednisolone dose following the OCS Optimization Phase. Maintenance (MN) dose was the mean of all daily prednisone/prednisolone doses during the MN Phase (weeks 20 to 24). The percent reduction of OCS dose during weeks 20 to 24 compared to BL dose was calculated as: 100 x (BL dose minus MN dose)/BL dose. Asthma control between weeks 20 and 24 was defined as no clinically significant exacerbation (worsening of asthma that required use of systemic corticosteroids or hospitalization and/or emergency department visits) during this period. Analysis was performed using a binary logistic regression model with terms for treatment group, region, duration of OCS use at BL (<5 years vs. >=5 years) and BL OCS dose.
Time Frame: Baseline; Weeks 20 to 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 66 | 69
Participants
  50 to 100% | 22 | 37
  <50% or no decrease/lack of asthma control/WD | 44 | 32

3. Secondary Outcome: Number of Participants Who Achieved a Reduction of Their Daily OCS Dose to <=5.0 mg During Weeks 20 to 24 While Maintaining Asthma Control
Description: Maintenance (MN) dose was the mean of all daily prednisone/prednisolone doses during the MN Phase (weeks 20 to 24). Asthma control between weeks 20 and 24 was defined as no clinically significant exacerbation (worsening of asthma that required use of systemic corticosteroids or hospitalization and/or emergency department visits) during this period. Number of participants who achieved a reduction of their daily OCS dose to <=5.0 mg was based on the value of the MN dose. Analysis was performed using a binary logistic regression model with terms for treatment group, region, duration of OCS use at BL (<5 years vs. >=5 years) and BL OCS dose.
Time Frame: Weeks 20 to 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 66 | 69
Participants
  <=5 mg/day | 21 | 37
  >5 mg/day or lack of asthma control or WD | 45 | 32

4. Secondary Outcome: Number of Participants Who Achieved a Total Reduction of OCS Dose During Weeks 20 to 24 While Maintaining Asthma Control
Description: MN dose was the mean of all daily prednisone/prednisolone doses during the MN Phase (weeks 20 to 24). Asthma control between weeks 20 and 24 was defined as no clinically significant exacerbation (worsening of asthma that required use of systemic corticosteroids or hospitalization and/or emergency department visits) during this period. The number of participants who achieved a total reduction of OCS dose was based on the value of the MN dose. Total reduction implied no OCS use during the entire MN phase. Analysis was performed using a binary logistic regression model with terms for treatment group, region, duration of OCS use at BL (<5 years vs. >=5 years) and BL OCS dose.
Time Frame: Weeks 20 to 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 66 | 69
Participants
  0 mg/day | 5 | 10
  OCS taken or lack of asthma control or WD | 61 | 59

5. Secondary Outcome: Median Percentage Change From Baseline in Daily OCS Dose During Weeks 20 to 24 While Maintaining Asthma Control
Description: BL dose was the prescribed optimized prednisone/prednisolone dose following the OCS Optimization Phase. MN dose was the mean of all daily prednisone/prednisolone doses during the MN Phase (weeks 20 to 24). The percent change of OCS dose during weeks 20 to 24 compared to BL dose was calculated as: 100 x (MN dose minus BL dose)/BL dose. Asthma control between weeks 20 and 24 was defined as no clinically significant exacerbation (worsening of asthma that required use of systemic corticosteroids or hospitalization and/or emergency department visits) during this period. For participants who withdrew from the study prior to the Maintenance Phase, and for participants with a lack of asthma control during the Maintenance Phase, a value equal to the minimum percent reduction in OCS use across all subjects was imputed for the analysis.
Time Frame: Baseline; Weeks 20 to 24
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Percentage reduction in OCS dose
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 66 | 69
Percentage reduction in OCS dose | 0.0 [-33.3 to 20.0] | -50.0 [-75.0 to -20.0]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were defined as events occurring from the first dose of investigational product until 28 days after the last dose of investigational product, up to 24 weeks.
Description: SAEs and Non-serious AEs were collected in members of Intent-to-Treat (ITT) Population, comprised of all participants who were randomized and who received at least one dose of study medication.
Arm/Group | Placebo | Mepolizumab 100 mg SC
Serious Adverse Events (participants affected / at risk) | 12/66 | 1/69
Other Adverse Events (participants affected / at risk) | 53/66 | 47/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | Mepolizumab 100 mg SC (N=69)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pneumonia (Infections and infestations) | 3 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Post gastric surgery syndrome (Injury, poisoning and procedural complications) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | Mepolizumab 100 mg SC (N=69)
Headache (Nervous system disorders) | 14 | 14
Nasopharyngitis (Infections and infestations) | 10 | 10
Bronchitis (Infections and infestations) | 6 | 7
Sinusitis (Infections and infestations) | 6 | 7
Fatigue (General disorders) | 4 | 7
Nausea (Gastrointestinal disorders) | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Adrenal insufficiency (Endocrine disorders) | 4 | 3
Pyrexia (General disorders) | 4 | 3
Injection site reaction (General disorders) | 2 | 4
Oedema peripheral (General disorders) | 2 | 4
Rhinitis (Infections and infestations) | 1 | 5
Dizziness (Nervous system disorders) | 3 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Hypersensitivity (Immune system disorders) | 3 | 1
Influenza (Infections and infestations) | 1 | 3
Injection related reaction (Injury, poisoning and procedural complications) | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Toothache (Gastrointestinal disorders) | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Cystitis (Infections and infestations) | 2 | 1
Otitis media (Infections and infestations) | 2 | 1
Sinus headache (Nervous system disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Eye pruritus (Eye disorders) | 2 | 0
Haematoma (Vascular disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Oral candidiasis (Infections and infestations) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Tooth infection (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.